CLINICAL TRIAL: NCT06177483
Title: Bioavailability Evaluation of a Micellar Curcumin Formulation (curQ+) Versus 95% Curcumin Extract in Healthy Individuals
Brief Title: Bioavailability Evaluation of CurQ+ Curcumin Formulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ESM-CLN#2023T02
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bioavailability
Keywords: Bioavailability, Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel group absorption study
Masking Description: Open label - all are aware of intervention assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 95% curcumin extract powder (Active Comparator): 1,265 mg of 95% curcumin extract (minimum 1,200 mg of curcuminoids) in three #0 vegetarian capsules as a single oral dose
  Interventions: Dietary Supplement: 95% curcumin extract powder
- curQ+ curcumin formulation (Experimental): 2,860 mg of curQ+® containing a total of 400 mg of curcuminoids in six #0 vegetarian capsules as a single oral dose
  Interventions: Dietary Supplement: curQ+ curcumin formulation

INTERVENTIONS:
Dietary Supplement: 95% curcumin extract powder — 95% curcumin extract powder
  Arms: 95% curcumin extract powder
Dietary Supplement: curQ+ curcumin formulation — curQ+ curcumin formulation
  Arms: curQ+ curcumin formulation

SUMMARY:
This study is intended to evaluate how significantly a proprietary curcumin formulation (curQ+®) results in greater bioavailability compared to 95% curcumin extract over a 6-hour time period following a single oral dose in healthy men & women.

DETAILED DESCRIPTION:
This study is intended to evaluate how significantly a proprietary curcumin formulation (curQ+®) results in greater bioavailability compared to 95% curcumin extract over a 6-hour time period following a single oral dose in healthy men & women. Bioavailability will be based upon producing the greatest plasma curcumin concentration (AUC). Secondarily, this study is intended to evaluate the safety and tolerability of the curQ+® curcumin formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects must be 18-75 years of age at the time of Screening.
2. Subjects must be willing to refrain from consuming the spice turmeric or any dietary supplements containing turmeric or curcumin (except for the study products) throughout the entire study and for 14 days prior to screening.
3. Subjects must be available for and willing to attend all evaluation visits.
4. Subjects must be able and willing to give informed consent.
5. Subjects participating in prior studies evaluating curQ+® or curcumin can participate in the present study so long as they are not currently taking a curcumin-containing supplement (including turmeric) and have not done so for 14 days prior to screening.

Exclusion Criteria:

1. Subject is currently receiving therapy with remission-inducing drugs (i.e. methotrexate, TNF biologics, etc.), immunosuppressive drugs (i.e. corticosteroids, transplantation medications, etc.).
2. Subjects must not have taken turmeric- or curcumin-containing dietary supplements within 14 days prior to screening evaluation.
3. Subject has been diagnosed with any clinically significant confounding metabolic disease or condition that would interfere with the study evaluation, as judged by the clinical investigator (slow or fast metabolism resulting from hypo- or hyper-thyroidism, Cushing's Syndrome, Diabetes (except for fully resolved gestational diabetes), etc.) or any conditions that would affect absorption in the GI tract (i.e. inflammatory bowel disease, celiac disease, Behçet's Syndrome, systemic sclerosis, etc.).
4. Subject has known allergy to any of the investigational products, including but not limited to turmeric, curcumin, coconut or coconut oil, and sunflower oil. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study.
5. Subject's body weight is greater than 300 pounds (136.1 kg) at the time of Screening.
6. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of the first baseline evaluation.
7. Pregnant and/or breastfeeding women, or women who intend to become pregnant during the course of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Absorption of curcumin | 6 hours
  difference between the absorption of curQ+ versus 95% curcumin powder

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Posey, PhD, Principal Investigator — UTHealth
Locations (1):
- University of Texas Health Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.